CLINICAL TRIAL: NCT01761422
Title: Myocardial Inflammation in Systemic Lupus Erythematosus
Status: Active, not recruiting | Type: Observational
Sponsor: Stacy Ardoin MD (Other)
Responsible Party: Sponsor-Investigator, Stacy Ardoin MD, Assistant Professor-Clinical, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2012H0132
Record Dates: First submitted 2013-01-03; First posted 2013-01-04 (Estimated); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: SLE

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- SLE active flare: Patients who are having an active flare of their lupus confirmed by labs

SUMMARY:
The goal is to assess for myocardial edema on cardiac MRI during SLE flare to assess for myocardial inflammation.

DETAILED DESCRIPTION:
The over-arching goal of this work is to further the understanding of myocardial damage in systemic lupus erythematosus (SLE) using state of the art CV imaging to investigate a novel potential mechanism of CV injury in SLE, subclinical myocardial inflammation.

Aim 1: Investigate an alternative pathway for CV morbidity in SLE by measuring myocardial edema at time of moderate to severe flare and compare values to post-flare studies and historical healthy controls.

Hypothesis 1: Myocardial edema, measured quantitatively with T2 CMR mapping during moderate to severe SLE flare will be significantly increased compared to 1) historical controls and 2) in SLE patients after resolution of flare.

Aim 2: Perform exploratory analyses investigating relationships between myocardial edema on CMR and markers of SLE disease activity and CV risk factors.

Hypothesis 2: Markers of disease activity including inflammatory makers (ESR and high sensitivity c-reactive protein), complement and autoantibody levels will predict the presence of T2 CMR detected myocardial edema during flare.

ELIGIBILITY:
Inclusion Criteria:

* • Diagnosis of SLE by American College of Rheumatology Classification Criteria [21]

  * Active SLE Flare defined by Systemic Lupus Erythematosus Disease Activity Index (SLEDAI)[22] > 6 or British Isles Lupus Assessment Group (BILAG) Index A or B.[23]

Exclusion Criteria:

* Pregnant
* Allergy to gadolinium
* Severe claustrophobia
* Renal replacement therapy or glomerular filtration rate (GFR) < 30 mL/min/1.75m²
* Medically unstable for transportation to Ross MRI scanner. Stability will be defined as: not on mechanical ventilation, HR < 120 BPM, MAP > 65 mmHg. The treating providers' input on the patient's stability will also be considered in addition to these criteria
* Weight > 500 pounds
* MR incompatible implanted devices such as neurostimulator pacemakers and implantable defibrillators, presence of intracranial metal or any metal not compatible with CMR

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults ages 18 years and older who are diagnosed with SLE
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2012-07-01; Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
T2 edema on Cardiac MRI | 3 months
  Compare T2 edema at flare and 3 months later

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Ardoin, MD, Principal Investigator — Ohio State University
Locations (1):
- Stacy Payne Ardoin, Columbus, Ohio, United States